CLINICAL TRIAL: NCT02553356
Title: A Single-Dose, Open-Label, Randomized, Food Effect Study in Healthy Volunteers With PT2385 Tablets
Brief Title: PT2385-102 Food Effect Study of PT2385 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peloton Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PT2385-102
Record Dates: First submitted 2015-09-11; First posted 2015-09-17 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Female Subjects
MeSH Terms: interventions — PT2385

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted (Experimental): PT2385 taken after fasting.
  Interventions: Drug: PT2385
- Non-Fasting (Experimental): PT2385 taken after eating a high calorie meal.
  Interventions: Drug: PT2385

INTERVENTIONS:
Drug: PT2385

SUMMARY:
This Phase 1, single-dose study will be conducted in adult female subjects (N = 16) who are in general good health and selected for participation in the study according to the selection criteria. This study will assess the effect of food on the pharmacokinetics of PT2385 Tablets. The study will consist of two periods and will be conducted in a crossover fashion.

DETAILED DESCRIPTION:
Subjects will be randomized in equal numbers to two sequences of meal conditions (fasting and non-fasting). Serial blood samples will be collected for after dose administration in each period. Subjects will be confined at the clinical research for a portion of each period.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 45 years of age;
* If of childbearing potential, willing to practice methods of birth control;
* If of childbearing potential, must be non-pregnant and non-lactating and have a negative serum pregnancy test result prior to enrollment into the trial;
* Has a body mass index (BMI) between 19 and 32 kg/m2;
* Willing and able to give written informed consent for study participation and provide consent for access to medical data;
* Willing and able to cooperate with all aspects of the protocol.

Exclusion Criteria:

* Any vaccination within 30 days before start of this study and throughout the study;
* Use of or need for any systemic drug(s) including vitamins or herbal preparations other than drugs used for contraception, within 30 days before entry into the study or during the study;
* Use of aspirin, non-steroidal anti-inflammatory agents, or acetaminophen within 5 days prior to the ingestion of the study drug;
* Donation or receipt of blood or blood components within the 4 weeks prior to the start of the study;
* Any diagnostic or intervention procedure requiring a contrast agent within the 30 days prior to the start of study participation;
* Abnormal blood pressure or pulse rate;
* Abnormal screening electrocardiogram (ECG);
* Use of tobacco or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.);
* Consumption of alcohol or xanthine-containing products;
* Consumption of grapefruit, star fruit, Seville oranges, or products containing any of these ingredients;
* Receipt of any investigational agent within 30 days;
* A positive history of drug abuse or a positive test result for drug(s) of abuse;
* Female subjects who are planning a pregnancy or are pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Effect of food on the pharmacokinetics of a single dose of PT2385 Tablets administered to normal healthy adult subjects (Cmax). | 6 days
  Peak Plasma Concentration (Cmax) will be assessed in both the fasting and non-fasting conditions and compared.

SECONDARY OUTCOMES:
Safety and tolerability of PT2385 Tablets in normal healthy adult subjects by reviewing the incidence of treatment-emergent adverse events. | 30 days
  Analyses will consist of data summaries for AEs/SAEs
Pharmacodynamic (PD) effects of treatment with PT2385 Tablets (plasma levels). | 6 days
  Variability in biomarkers will be correlated with plasma levels of PT2385.

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States